CLINICAL TRIAL: NCT03049046
Title: Protocol CC100B. CC100: Phase 1 Multiple-Dose Safety and Tolerability in Subjects With ALS
Brief Title: CC100: Phase 1 Multiple-Dose Safety and Tolerability in Subjects With ALS
Acronym: CC100B
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chemigen, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CC100B; 1R01FD004790-01A2 (FDA)
Record Dates: First submitted 2017-02-03; First posted 2017-02-09 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CC100 250 mg (Active Comparator): CC100 250 mg once daily by mouth for 7 days
  Interventions: Drug: CC100
- CC100 500 mg (Active Comparator): CC100 500 mg once daily by mouth for 7 days
  Interventions: Drug: CC100
- CC100 1000 mg (Active Comparator): CC100 1000 mg once daily by mouth for 7 days
  Interventions: Drug: CC100
- Placebo (Placebo Comparator): Placebo once daily by mouth for 7 days
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: CC100 — synthetic caffeic acid phenethylester
  Other Names: synthetic caffeic acid phenethylester
  Arms: CC100 1000 mg; CC100 250 mg; CC100 500 mg
Drug: Placebos — Diluent
  Other Names: Placebo oral liquid
  Arms: Placebo

SUMMARY:
Approximately 21 subjects with amyotrophic lateral sclerosis (ALS) will be randomized (6 to 1) to receive by mouth seven morning doses of CC100 or placebo for 7 days. Subjects are required to stay in the Clinic for approximately 9 hours following the first and last dose. Subjects will also have a mid-week clinic visit and will be contacted by phone within 3 to 5 days after the last dose.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
Primary objective: to assess the safety and tolerability of multiple doses of orally administered CC100 in subjects with amyotrophic lateral sclerosis (ALS). Secondary objectives: to determine pharmacokinetics and pharmacodynamics of CC100 in plasma after single and after multiple doses; and to determine short-term effects of CC100 on potential blood-cell ALS biomarkers.

Study Design: Phase 1 double-blind, randomized, placebo-controlled multiple-dose of three CC100-dose cohorts. Approximately 18 subjects will receive CC100. Approximately 3 subjects will be randomized to placebo (across 3 cohorts). Periodic Assessment Committee safety reviews. Note: Participation will not exclude subjects from future CC100 studies Criteria for Evaluation: Safety Endpoints: Adverse events, blood chemistry, hematology, urinalysis, vital signs, 12-lead ECGs. Pharmacokinetic (PK)/Pharmacodynamic (PD): Plasma for CC100 concentrations (PK). Blood collected at baseline and after each subject's last dose will be assayed for potential biomarker(s). Stored specimens will be de-identified or combined for validating diagnostic tools/assays related to ALS. Statistical Methods: A minimum of 6 subjects per CC100 dose group and 3 placebo-dosed subjects (total across cohorts) are considered sufficient to evaluate initial safety and tolerability for the cohorts. Pharmacokinetic parameter estimates will be calculated by standard noncompartmental methods of analysis. Absolute bioavailability of administration will be estimated based on the total area under the time- concentration curve (AUC0-∞).

ELIGIBILITY:
Inclusion Criteria:

* Have definite or probable ALS with a forced vital capacity of >60% predicted.
* Men must practice a reliable method of birth control during study and for 2 weeks following study. Women must be non-fertile or post-menopausal.
* Riluzole is allowed if dose has been stable for at least 30 days. Other allowed medications: lipid-lowering drugs, anti-hypertensives, anti-depressants, oral medications for type II diabetes, estrogen replacement therapy, thyroid replacement therapy, antihistamines, antacids, nonsteroidal anti-inflammatory drugs (except indomethacin), histamine H2-receptor antagonists, proton-pump inhibitors, calcium supplements, topical eye medications, and topical antibiotics.

Exclusion Criteria:

* Greater than 250 pounds
* Have serious or unstable illnesses as determine by the investigator.
* Have current or a history of asthma or severe drug allergies or pollen allergy.
* Have had serious infectious disease affecting the brain within the preceding 5 years; or have existing evidence of serious infection.
* Have laboratory test values that are considered clinically significant as determined by the investigators.
* Have ECG abnormalities that are clinically significant.
* Have donated blood (a pint or more) or received an experimental drug within 30 days prior to dosing.
* Have a history of chronic alcohol or drug abuse within the past 2 years.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2017-04-07 (Actual); Primary Completion 2018-01-30 (Estimated); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability: Adverse events, safety labs, vital signs, and ECGs | From start of first dose to a minimum of 3 days after last dose
  Safety and tolerability assessed by group/dose measured by number of unsolicited adverse events (MedDRA), and changes in blood chemistry, hematology, urinalysis, vital signs, and 12-lead ECGs from baseline (prior to dosing).

SECONDARY OUTCOMES:
Pharmacokinetics (PK)--Peak plasma concentration (Cmax) | 0.5, 1, 2, 4, and 8 hours after first and last dose
  Cmax after first (single) and last (multiple) CC100 doses
Pharmacokinetics (PK)--Area under the plasma concentration versus time curve (AUC) | 0.5, 1, 2, 4, and 8 hours after first and last dose
  AUC after first (single) and last (multiple) CC100 doses
Pharmacokinetics (PK)--Half life (T 1/2) | 0.5, 1, 2, 4, and 8 hours after first and last dose
  Estimated half-life after first (single) and last (multiple) CC100 doses
Pharmacodynamics (PD)--Monocyte chemotactic protein 1 (MCP-1) | Pretreatment and 8 hours post last dose
  Short-term effects of CC100 on potential ALS inflammation biomarker MCP-1
Pharmacodynamics (PD)--Excitotoxicity/oxidative stress biomarkers | Pretreatment and 8 hours post last dose
  Short-term effects of CC100 on potential ALS excitotoxicity/oxidative stress biomarkers: Heme oxygenase-1 (HMOX-1)/thioredoxin (TRX)/heat-shock protein 70 (HSP-70)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, IU Health Physicians Neurology, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Single-site study

REFERENCES:
- [Derived] Chang GJ, Yeh YH, Chen WJ, Hsu SC, Lai YJ, Chang CJ, Lee HY. Caffeic Acid Phenethyl Ester Improves Right Ventricular Function and Reduces Arrhythmogenesis by Attenuating Structural and Electromechanical Remodeling in Pulmonary Arterial Hypertensive Rats. Phytother Res. 2026 Jan 26. doi: 10.1002/ptr.70219. Online ahead of print. PMID 41587816